CLINICAL TRIAL: NCT00846911
Title: AVANTI - Avelox® in Acute Exacerbations of Chronic Bronchitis
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Global Medical Affairs Head, Bayer HealthCare AG
Other Study IDs: 14689; AX0701 (Other: Company Internal); 13598 (Other: Company Internal); 13855 (Other: Company Internal); 13856 (Other: Company Internal); 13857 (Other: Company Internal); 14008 (Other: Company Internal); 14007 (Other: Company Internal); 14009 (Other: Company Internal)
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Bronchitis, Chronic
Keywords: Acute Exacerbation of Chronic Bronchitis (AECB) patients
MeSH Terms: conditions — Bronchitis, Chronic | interventions — Moxifloxacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — Patients with acute exacerbation of chronic bronchitis for whom the physician decided to prescribe moxifloxacin

SUMMARY:
The objective of this global non-interventional study is to evaluate the impact of Acute Exacerbation of Chronic Bronchitis(AECB) on the patient and the community as well as the safety and effect of a treatment with Moxifloxacin tablets in daily life clinical practice. This includes data on the course of symptom relief, speed of return to normal daily life activities as well as records on adverse events.

This study will be performed in accordance with international guidelines like EMEA (EMEA, EUDRALEX Volume 9A, Pharmacovigilance for Medicinal Products for Human Use) as well as local laws.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 35 years of age with a diagnosis of Acute Exacerbation of Chronic Bronchitis (AECB) and decision taken by the investigator to treat with Avelox.

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 2672 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Time until improvement of acute exacerbation | End of study

SECONDARY OUTCOMES:
Time until cure of acute exacerbation | End of study
Severity of AECB according to Antonisen criteria | Baseline
Impact of AECB on daily life activities | Baseline
Safety of Avelox under daily life treatment conditions | Throughout treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (8):
- Many Locations, Albania
- Many Locations, Bosnia and Herzegovina
- Many Locations, Kazakhstan
- Many Locations, Moldova
- Many Locations, North Macedonia
- Many Locations, Russia
- Many Locations, Slovakia
- Many Locations, Ukraine

REFERENCES:
- [Derived] Chuchalin A, Zakharova M, Dokic D, Tokic M, Marschall HP, Petri T. Efficacy and safety of moxifloxacin in acute exacerbations of chronic bronchitis: a prospective, multicenter, observational study (AVANTI). BMC Pulm Med. 2013 Jan 23;13:5. doi: 10.1186/1471-2466-13-5. PMID 23343427